CLINICAL TRIAL: NCT06914518
Title: Polynucleotide and Hyaluronic Acid-based Gel as Adjunctive Therapy to Non- Surgical Treatment of Intraosseous Peri-implant Defect. A 6-month Randomized Clinical Trial
Brief Title: Polynucleotide and Hyaluronic Acid-based Gel as Adjunctive Therapy to Non- Surgical Treatment of Intraosseous Peri-implant Defect. A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER-ECL-2023-06
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Peri-implantitis
Keywords: peri-implantitis; non-surgical treatment; non-surgical treatment per-implantitis; hyaluronic acid
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- non-surgical therapy (Active Comparator): Standardized peri-implant non-surgical therapy will be performed as follows: local anaesthesia (articaine 4% and adrenaline 1:100,000), debridement of the implant surfaces with ultrasonic devices (Newtron P5, Satelec Acteon; Olliergues, France) with the H3 dental ultrasonic scaler (H3, Satelec Acteon; Olliergues, France), curettage of the bone defect (SyG 7/89 Everdge, Hu-Friedy; Chicago, IL, USA) and supra- and submucosally cleaning using an air polisher with sub- gingival tip (EMS Air-flow® with erythritol-based powder containing)
  Interventions: Procedure: Non-Surgical Intervention
- Test group: adjunctive PN-HA gel (Experimental): Standardized peri-implant non.surgical therapy will be performed as follows: local anaesthesia (articaine 4% and adrenaline 1:100,000), debridement of the implant surfaces with ultrasonic devices (Newtron P5, Satelec Acteon; Olliergues, France) with the H3 dental ultrasonic scaler (H3, Satelec Acteon; Olliergues, France), curettage of the bone defect (SyG 7/89 Everdge, Hu-Friedy; Chicago, IL, USA) and supra- and submucosally cleaning using an air polisher with sub- gingival tip (EMS Air-flow® with erythritol-based powder containing). At the end of the peri-implant non-surgical therapy a viscoelastic gel containing a fixed combination of natural origin PN (10 mg/ml, 1%) and HA with molecular weight > 1500 kDa (10 mg/ml, 1%) (REGENFASTe, Mastelli S.r.l., Sanremo, Italy) will be injected in the peri-implant sulcus.
  Interventions: Other: viscoelastic gel containing a fixed combination of natural origin PN (10 mg/ml, 1%) and HA with molecular weight > 1500 kDa (10 mg/ml, 1%); Procedure: Non-Surgical Intervention

INTERVENTIONS:
Other: viscoelastic gel containing a fixed combination of natural origin PN (10 mg/ml, 1%) and HA with molecular weight > 1500 kDa (10 mg/ml, 1%) — At the end of the standardized peri-implant non-surgical therapy a viscoelastic gel containing a fixed combination of natural origin PN (10 mg/ml, 1%) and HA with molecular weight > 1500 kDa (10 mg/ml, 1%) (REGENFASTe, Mastelli S.r.l., Sanremo, Italy) will be injected in the peri-implant sulcus.
  Arms: Test group: adjunctive PN-HA gel
Procedure: Non-Surgical Intervention — Standardized peri-implant non-surgical therapy will be performed as follows: local anaesthesia (articaine 4% and adrenaline 1:100,000), debridement of the implant surfaces with ultrasonic devices (Newtron P5, Satelec Acteon; Olliergues, France) with the H3 dental ultrasonic scaler (H3, Satelec Acteon; Olliergues, France), curettage of the bone defect (SyG 7/89 Everdge, Hu-Friedy; Chicago, IL, USA) and supra- and submucosally cleaning using an air polisher with sub- gingival tip (EMS Air-flow® with erythritol-based powder containing

SUMMARY:
This randomized, placebo-controlled clinical trial evaluates the efficacy of a polynucleotide and hyaluronic acid-based gel (PN-HA) as adjunctive therapy to non-surgical flapless treatment of peri-implantitis. The main goal is to assess probing pocket depth (PPD) reduction after 6 months compared to placebo.

Study Design:

* Type: Interventional (Clinical Trial)
* Allocation: Randomized (computer-generated blocks)
* Intervention Model: Parallel assignment
* Masking: Single-blind (examiner-blinded)
* Primary Purpose: Treatment
* Estimated Enrollment: 32 participants
* Duration: 6 month follow-up

DETAILED DESCRIPTION:
Study design This study will be a randomized controlled, clinical trial with 6 months follow-up.

Participants:

Subjects eligible for the study will be identified from patients referred to the Clínica Universitària d'Odontologia - UIC Barcelona at the Periodontology Department. All study subjects will provide written informed consent before participating in the study.

Inclusion criteria: ≥18 years old, ≥1 implant with peri-implantitis and intraosseous defect ≥3mm, good oral hygiene, modifiable prosthesis.

Exclusion criteria: systemic diseases, pregnancy, recent antibiotic use, smoking >10 cigarettes/day, poor plaque control, implant mobility.

Interventions:

One week prior to submucosal debridement, all patients will receive professional supragingival teeth/implant prophylaxis, oral hygiene instructions, and implant-supported prosthesis corrections if needed to provide an oral environment favourable to wound healing. All subjects will receive a session of full-mouth professional prophylaxis, including scaling and tooth polishing. Supragingival and supramucosal debridement by means of an ultrasonic device (DTE-D5, Woodpecker®, Guilin, China) using a plastic tip (Hu-Friedy®, Rockwell St, Chicago, IL, USA) will be performed. Finally, the prosthetic components will be polished using a rubber cup.

Additionally, when implant-supported prosthesis does not allow access for proper oral hygiene, prosthesis corrections will be performed according to the protocol described by de Tapia et al. (2019)

Individualized instructions in proper oral hygiene measures will be given to all patients enrolled in the study

Control Group: Non-surgical peri-implant debridement without adjunctive gel.

Test Group: Same treatment plus application of a viscoelastic gel containing a fixed combination of natural origin PN (10 mg/ml, 1%) and HA with a molecular weight > 1500 kDa (10 mg/ml, 1%) (REGENFAST®, Mastelli S.r.l., Sanremo, Italy) injected into the peri-implant sulcus.

All patients undergo professional hygiene and oral hygiene instruction. Non-surgical treatment includes ultrasonic and air-polishing debridement, with or without PN-HA gel application.

Follow-Up Schedule:

Baseline (T0): clinical, radiographic, biochemical, mmicrobilogical assessment and PROMS collections.

Follow-up:

Day 14: Microbiological and biochemical parameters, PROMS Month 3, 6: clinical/radiographic reassessment and maintenance

Data collection A guidebook will be prepared to standardize procedures throughout the protocol, step by step, for all questionnaires and evidence collection. The data will be transferred to a computerized database.The study variables will be recorded in a case report form (CRF) specially designed for the study. Each study patient will be assigned a numerical code comprising a 3-digit patient code.

Anthropometric and sociodemographic data An interview will be conducted to obtain information regarding age, race, gender, medical history, medication, and health behaviour (smoking habit). Smoking behaviour will be specified as 3 categories: never-smoker (i.e., < 100 cigarettes per lifetime), former smoker, or current smoker (light smokers: < 10 cigarettes/day). Patients will be asked about their tobacco smoke exposure in terms of consumption (i.e. the number of cigarettes consumed per day); duration (i.e. the number of years of smoking); and lifetime exposure (i.e. pack-years) (34). In case of former smokers, patients will be asked about the time since smoking cessation.

Clinical measurements A single calibrated examiner (M.I.A.) will assess the following clinical parameters at baseline (i.e., submucosal debridement), 3 and 6 months after the therapy using a periodontal probe (PCP-UNC 15; Hu-Friedy, Chicago, IL, USA).

At the implant level, in six sites around each implant, the following clinical variables will be recorded:

1. Modified plaque index (mPI) .
2. Modified Plaque Index (mPI) is a dental plaque scale as follows 0 = No plaque, 1 = Separate flecks of plaque at the cervical margin;2 = Plaque can be seen by naked eye.3 = Abundance of soft matter. The lower the number the less plaque is present on the tooth.
3. Modified bleeding index (mBI). This variable will be dichotomized in presence/absence of bleeding on probing (BoP) 0=No bleeding when a periodontal probe is passed along the mucosal margin adjacent to the implant, 1= Isolated bleeding spots visible, 2= Blood forms a confluent red line on mucosal margin, 3= Heavy or profuse bleeding
4. Suppuration (SUP) on probing: presence or absence of suppuration after gentle probing
5. Peri-implant pocket depth (PPD): distance (mm) from the mucosal margin to the base of the probable pocket.
6. Bleeding on porbing (BoP) will be assessed dichotomously in six sites per implant.
7. Keratinized mucosa width (KMW) will be measured as the distance (mm) from the mucosal margin to the mucogingival junction at the mid-buccal aspect of the implant with the resin splint.

Moreover, at the patient level, the following variables will be assessed at baseline and at 3 and 6 months after the therapy:

Full-mouth plaque index (FMPI) assessed dichotomously at four sites per tooth (mesial, buccal, lingual, distal). Presence or absence will be recorded after staining with an erythrosine disclosing dye (Plac-Control®, Dentaid SL, Cerdanyola, Spain). Presence of plaque will be scored if an area of clearly stained material is present along the gingival margin and if the material can be removed with the side of the probe. The percentage of surfaces with plaque out of the total number of examined tooth surfaces will be calculated (37).

Full-mouth bleeding index (FMBI) assessed dichotomously as presence or absence of bleeding after 30 seconds of gently probing. The proportion of bleeding surfaces out of the total number of examined surfaces will be calculated (38).

Furthermore, implant position (maxilla/mandible and incisors, canines, premolars, and molars) and implant system will be further recorded as well as the type of prosthesis (cemented/screw- retained).

In case patients have more than one implant, all the implants will be treated but only the implant with the most severe condition will be included in the study (i.e., the implant with the deepest PPD at baseline).

Radiographic assessment

Intra-oral periapical radiographs with a bite block will be taken using the long cone paralleling technique (7mA- 60kV/20ms) at baseline and at 3 and 6 after the peri-implant therapy. A film holder will be modified by placing a registration material (Optosil®) on the bite blocks to index the dentition and using a paralleling cone technique. Then, reproducible measurements at each examination time point will be obtained. The digitally obtained X-rays will be transferred into a software program (Image J; NIH, Bethesda, MD, USA) and calibrated using the known implant dimensions (i.e., diameter or length) as reference values. The following measurements will be recorded by a blinded and calibrated examiner at the mesial and distal aspects of the treated implants:

* Bone level (BL): distance (mm) between the implant shoulder and the base of the defect.
* Intra-bony defect (ID): distance (mm) between the bottom of the defect and the line connecting the distal and mesial interproximal bone crest.
* Intra-bony defect width (WD): distance (mm) between the distal and mesial interproximal bone crest and the implant surface.
* Angulation of the intra-bony defect (AD): angle resulted from a vertical line along the outer implant surface and a line extending along the peri-implant bone defect.

Laboratory analyses Enzyme-linked immunosorbent assay (ELISA) PICF samples will be taken in each implant at the deepest PPD site at baseline, and 14 days, 3 and 6 months after the treatment. The area will be isolated with cotton rolls and gentle cleaning with air and a gauze to remove supragingival plaque deposits and potential saliva contamination. A paper strip of standard length and height (Periopaper®, Oraflow, Hewlett, NY, USA) will be inserted into the peri-implant pocket until mild resistance and will be felt and left in place for 30 s. Strips visually contaminated with blood will be discarded. Strips will be immediately placed in separate microcentrifuge tubes containing 250 ml phosphate- buffered saline and protease inhibitor cocktail (Sigma-Aldrich, Saint Louis, Missouri, USA). The samples will be immediately stored at -80 C until their biochemical analysis. Serum levels of IL-1β, IL-8, and TNF-α will be measured by a quantitative enzyme immunoassay technique, by using the Quantikine ELISA Kit according to the manufacturer's instructions (R & D System, Minneapolis, USA).

Quantitative polymerase chain reaction (q-PCR) Immediately after biochemical analysis, microbiological testing will be performed in the deepest peri-implant pocket of each subject at baseline, 14 days, 3 and 6 after the therapy. Following elimination of the supragingival biofilm, samples will be taken with two consecutive sterile medium paper points (Maillefer, Ballaigues, Switzerland). The paper points will be kept in place for 10 s and transferred into one empty sterilized 1.5 ml Eppendorf tube. A commercially available microbiological test (Dentaid®, Cerdanyola del Vallès, Barcelona) will be used. Presence and numbers of Aggregatibacter actinomycetemcomitans, Porhyromonas gingivalis, Prevotella intermedia, Tannerella forsythia, Parvimonas micra, Fusobacterium nucleatum, Campylobacter rectus and Treponema denticola will be determined (log CFU ml1). Microbial samples will be analyzed using quantitative polymerase chain reaction.

Patient-reported outcomes Patients of the test and control groups will be subjected to the 14-items oral health-related quality of life (OHIP-14sp) questionnaire in the Spanish version at the baseline and after 14 days as well as 6 months of follow-up (43) . Pain of the patients at baseline will be assessed using a visual analogue scale (VAS score; VAS 0-100, 100 reflecting the highest morbidity). Immediately after non-surgical therapy and after 14 days, will be assessed using a visual analogue scale (VAS score; VAS 0-100, 100 reflecting the highest morbidity). Medication consumption and spontaneous bleeding, pain and swelling in the two-weeks following therapy will be assessed.

Randomization:

Subjects will be randomly assigned by a computer-generated table to receive one of the two treatments. A balanced random permuted block approach (4-unit block size) will be used to prepare the randomization gel (PN-HA (test) or placebo (control)) to avoid unequal balance between treatments.

Outcome Measures:

Primary:

PPD reduction at 3 and 6 months.

Secondary:

Clinical: mPI, BoP, mBI, SoP, keratinized mucosa width Radiographic: marginal bone level, defect width and angulation Microbiological: presence of selected pathogens via qPCR Biomarkers: IL-1β, IL-8, TNF-α in PICF (ELISA) PROMs: OHIP-14 questionnaire, VAS score, medication use

Examiners: blinding and calibration. All clinical evaluations will be performed by one investigator (M.I.A.), blinded concerning treatment modality. All radiological assessments will be performed by one investigator (M.C.S.), blinded concerning treatment modality. For validation, the radiographs of 20 patients will be randomly selected and remeasured to calculate the intra-examiner agreement. The same measurements will be calculated by another investigator (C.V.V.) and inter-examiner will be calculated.

Withdrawal of consent The Patient Information Sheet will clearly state that the patient can withdraw from the study at any time without prejudice or explanation. Such withdrawal will be documented in the medical record file. Losses to follow-up are taken into account in the sample size calculations (10%).

Statistical Analysis:

Sample size:

Sample size will be obtained from a comparable study on periimplantitis where the sample size was calculated according to their preliminary data. The test group showed a standard deviation (SD) of 1.703 mm and the control group of 1.803 mm with a mean difference of 1.214 mm, thus a sample of 32 patients, 16 per group, was estimated to provide 80% power with an α of .05, accounting for 10% attrition.

The patient will be considered the unit of analysis. To describe the qualitative variables, absolute frequencies, and percentages will be used. The description of quantitative variables will be performed using the mean, standard deviation (SD), median, and quartiles. A final model will be developed using back stepwise linear regression analysis including PPD as a dependent variable. The SPSS version 23.00 software (SPSS Inc., Chicago, IL, USA) will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

Subjects with (I) ≥ 18 years of age, the presence of at least one implant diagnosed with peri-implantitis, intraosseous ≥ 3mm defects, presence of screw-retained single-unit crowns and partial dental prosthesis that allowed correct access for brushing; and, if not, prostheses that could be modified.

Exclusion Criteria:

Subjects will be excluded from the study if they had received previous non-surgical peri-implantitis treatment during the last 6 months or surgical treatment, were pregnant or breast-feeding, had received antibiotic treatment in the previous 3 months, had systemic conditions that contraindicated treatment, smoking more than 10 cigarettes/day or presents a poor plaque control (Plaque Index < 20%), implant mobility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth | Baseline , 3 months, 6 months
  Peri-implant pocket depth: distance (mm) from the mucosal margin to the base of the probable pocket.

SECONDARY OUTCOMES:
Modified plaque index | Baseline , 3 months, 6 months
  Modified Plaque Index (mPI) is a dental plaque scale as follows 0 = No plaque, 1 = Separate flecks of plaque at the cervical margin;2 = Plaque can be seen by naked eye.3 = Abundance of soft matter. The lower the number the less plaque is present on the tooth.
Modified bleeding index | Baseline , 3 months, 6 months
  This variable will be dichotomized in presence/absence of bleeding on probing (BoP) 0=No bleeding when a periodontal probe is passed along the mucosal margin adjacent to the implant, 1= Isolated bleeding spots visible, 2= Blood forms a confluent red line on mucosal margin, 3= Heavy or profuse bleeding
Bleeding on porbing | Baseline , 3 months, 6 months
  Bleeding on porbing will be assessed dichotomously in six sites per implant
Keratinized mucosa width | Baseline , 3 months, 6 months
  Keratinized mucosa width (mm) will be measured as the distance (mm) from the mucosal margin to the mucogingival junction at the mid-buccal aspect of the implant with the resin splint.
Bone level | Baseline , 3 months, 6 months
  Radiographic distance (mm) between the implant shoulder and the base of the defect.
Intra-bony defect width | Baseline , 3 months, 6 months
  radiographic istance (mm) between the distal and mesial interproximal bone crest and the implant surface.
Angulation of the intra-bony defect | Baseline , 3 months, 6 months
  radiographic measurement of the angle resulted from a vertical line along the outer implant surface and a line extending along the peri-implant bone defect.
Serum levels of IL-1β, IL-8, and TNF-α | Baseline , 14 days
  Serum levels of IL-1β, IL-8, and TNF-α will be measured by a quantitative enzyme immunoassay technique, by using the Quantikine ELISA Kit according to the manufacturer's instructions (R & D System, Minneapolis, USA) (42).
Presence and numbers of Aggregatibacter actinomycetemcomitans, Porhyromonas gingivalis, Prevotella intermedia, Tannerella forsythia, Parvimonas micra, Fusobacterium nucleatum, Campylobacter rectus and Treponema denticola | Baseline , 14 days
  Samples will be taken with two consecutive sterile medium paper points (Maillefer, Ballaigues, Switzerland). The paper points will be kept in peri-implant sulcus for 10 s and transferred into one empty sterilized 1.5 ml Eppendorf tube.Presence and numbers of Aggregatibacter actinomycetemcomitans, Porhyromonas gingivalis, Prevotella intermedia, Tannerella forsythia, Parvimonas micra, Fusobacterium nucleatum, Campylobacter rectus and Treponema denticola will be determined (log CFU ml1). Microbial samples will be analyzed using quantitative polymerase chain reaction
Pain of the patients | baseline, after non surgical therapy, 14 days.
  Pain of the patients at baseline will be assessed using a visual analogue scale (VAS score; VAS 0-100, 100 reflecting the highest morbidity).

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Valles, Dentistry, Principal Investigator — Department of Periodontology, Universitat Internacional de Catalunya
Locations (2):
- Spain (2):
  - Clinica Universitaria ́̀ d'Odontologia - UIC Barcelona at the Periodontology Department, Sant Cugat del Vallès, Barcelona
  - 08195, Sant Cugat del Vallès, Bracelona

IPD SHARING:
Plan to Share IPD: No
privacy concerns and lack of explicit consent for secondary data use further limit the possibility of data sharing

REFERENCES:
- [Background] Asparuhova MB, Kiryak D, Eliezer M, Mihov D, Sculean A. Activity of two hyaluronan preparations on primary human oral fibroblasts. J Periodontal Res. 2019 Feb;54(1):33-45. doi: 10.1111/jre.12602. Epub 2018 Sep 27. PMID 30264516
- [Background] Rams TE, Degener JE, van Winkelhoff AJ. Antibiotic resistance in human chronic periodontitis microbiota. J Periodontol. 2014 Jan;85(1):160-9. doi: 10.1902/jop.2013.130142. Epub 2013 May 20. PMID 23688097
- [Background] Pilloni A, Schmidlin PR, Sahrmann P, Sculean A, Rojas MA. Effectiveness of adjunctive hyaluronic acid application in coronally advanced flap in Miller class I single gingival recession sites: a randomized controlled clinical trial. Clin Oral Investig. 2019 Mar;23(3):1133-1141. doi: 10.1007/s00784-018-2537-4. Epub 2018 Jun 30. PMID 29961138
- [Background] Blanco C, Pico A, Dopico J, Gandara P, Blanco J, Linares A. Adjunctive benefits of systemic metronidazole on non-surgical treatment of peri-implantitis. A randomized placebo-controlled clinical trial. J Clin Periodontol. 2022 Jan;49(1):15-27. doi: 10.1111/jcpe.13564. Epub 2021 Oct 28. PMID 34713471
- [Background] Nart J, Pons R, Valles C, Esmatges A, Sanz-Martin I, Monje A. Non-surgical therapeutic outcomes of peri-implantitis: 12-month results. Clin Oral Investig. 2020 Feb;24(2):675-682. doi: 10.1007/s00784-019-02943-8. Epub 2019 May 23. PMID 31123873
- [Background] Linares A, Sanz-Sanchez I, Dopico J, Molina A, Blanco J, Montero E. Efficacy of adjunctive measures in the non-surgical treatment of peri-implantitis: A systematic review. J Clin Periodontol. 2023 Jun;50 Suppl 26:224-243. doi: 10.1111/jcpe.13821. Epub 2023 May 4. PMID 37143407
- [Background] Linares A, Pico A, Blanco C, Blanco J. Adjunctive Systemic Metronidazole to Nonsurgical Therapy of Peri-implantitis with Intrabony Defects: A Retrospective Case Series Study. Int J Oral Maxillofac Implants. 2019 Sep/Oct;34(5):1237-1245. doi: 10.11607/jomi.7343. PMID 31528867